CLINICAL TRIAL: NCT01714752
Title: Evaluation of Left Ventricular Filling Pressures During Exercise: Comparative Study, Catheterization Versus Echocardiography
Brief Title: Evaluation of Left Ventricular Filling Pressures During Exercise
Acronym: PREFFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: French Federation of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-02
Record Dates: First submitted 2012-10-19; First posted 2012-10-26 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF); Left Ventricular End Diastolic Pressure (LVEDP)
Keywords: Diagnosis; Left ventricular end diastolic pressure (LVEDP); Exercise echocardiography; Left atrial remodeling
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise (Experimental): Patients perform exercise and pression measure is performed
  Interventions: Procedure: measure of left ventricular and diastolic pressure at exercise

INTERVENTIONS:
Procedure: measure of left ventricular and diastolic pressure at exercise

SUMMARY:
Heart failure with preserved ejection fraction (HFPEF) is common and is a real public health issue. Diagnosis, especially when there are no congestive signs, is difficult. It has been shown that many patients with suspected HFPEF had left ventricular (LV) filling pressures elevated only at exercise (normal at rest).

Using stress echocardiography and taking into account left atrial (LA) remodeling at rest as a "memory" of chronic elevation of filling pressures. We believe that it is possible to improve the noninvasive diagnosis of exercise elevation of the LV end-diastolic pressure (LVEDP).

DETAILED DESCRIPTION:
Purpose Heart failure with preserved ejection fraction (HFPEF) is common and is a real public health issue. Diagnosis, especially when there are no congestive signs, is difficult. It has been shown that many patients with suspected HFPEF had left ventricular (LV) filling pressures elevated only at exercise (normal at rest).

Hypothesis Using stress echocardiography and taking into account left atrial (LA) remodeling at rest as a "memory" of chronic elevation of filling pressures. We believe that it is possible to improve the noninvasive diagnosis of exercise elevation of the LV end-diastolic pressure (LVEDP).

Methods Prospective, monocentric and comparative study: catheterization versus echocardiography.

60 patients referred for coronary angiography will be recruited consecutively during their hospitalization.

Patients should perform a low intensity and short duration exercise, in both catheterization and echo labs (pedaling 3 minutes at 25Watts then, 3 minutes at 50W) The LVEDP will be measured invasively with a pigtail, at rest and at both levels of exercise.

Echocardiography will be performed within 24 hours after catheterization, after a full examination at rest, an identical exercise (same intensity, same duration, same position of the patient) than made in catheterization lab will be done. Following parameters will be recorded at both stress levels: trans mitral flow, mitral annular pulsed tissue Doppler imaging (both lateral and septal) and tricuspid regurgitation flow.

The doctor who will perform the echocardiographic acquisitions will not be informed of the results of catheterization. The acquisitions will be analyzed in a second time still blinded to the catheterization data.

The following echocardiographic parameters will be collected and compared to the invasive measurement of LVEDP:

* Ratio between pulsed Doppler peak E velocity and peak Ea velocity obtained with tissue Doppler imaging (E/Ea ratio) at rest and exercise,
* maximal LA volume indexed to body area
* (maximal LA volume) to (maximal LV volume) ratio.
* LA distensibility defined by: (maximal LA volume - minimal LA volume) / (minimal LA volume)
* LA Global longitudinal strain Finally, it will be investigated whether the combined use of E/Ea ratio at exercise with LA remodeling indices (of morphology and/or function) improves the performance characteristics of diagnostic test, compared to a separate use of these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for coronary angiography
* Sinus Rhythm
* Left ventricular Ejection Fraction > 50%

Exclusion Criteria:

* Age < 18years
* Hypertrophic Cardiomyopathy
* Cardiac transplantation
* Mitral stenosis
* Mitral insufficiency >2/4
* Severe calcification of mitral annulus
* Mitral prothesis or mitral repair
* aortic prothesis
* Severe aortic stenosis
* Atrial fibrillation
* Acute coronary syndrom < 3 months
* Left ventricular thrombus
* Severe renal Failure
* failure of radial way for coronary angiography
* coronary lesion indicating an angioplasty
* impossibility to perform an exercise
* refusal or inability to sign informed consent
* no French medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
E/Ea ratio | Day 1
  E/Ea ratio as a non-invasive index of Left Ventricular and diastolic pressure (LVEDP) at exercise

SECONDARY OUTCOMES:
left atrial (LA) morphology | Day 1
  To evaluate left atrial (LA) morphology at rest (maximal LA volume indexed to body area, maximal LA volume to maximal LV volume ratio) as an index of Left Ventricular end diastolic pressure (LVEDP) at exercise.
LA function at rest | Day 1
  To evaluate LA function at rest (distensibility, global longitudinal strain) as an index of Left Ventricular end diastolic pressure (LVEDP) at exercise.
E/Ea ratio at exercise with LA remodeling indices at rest | Day 1
  To investigate whether the combined use of E/Ea ratio at exercise with LA remodeling indices at rest (of morphology and/or function) improves the performance characteristics of diagnostic test compared to a separate use of these parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Nadjib Hammoudi, MD, Principal Investigator — Cardiology department - Pitié Salpêtrière Hospital
Locations (1):
- Pitié Salpêtrière Hospital - Cardiology Department, Paris, France

REFERENCES:
- [Derived] Hammoudi N, Laveau F, Helft G, Cozic N, Barthelemy O, Ceccaldi A, Petroni T, Berman E, Komajda M, Michel PL, Mallet A, Le Feuvre C, Isnard R. Low level exercise echocardiography helps diagnose early stage heart failure with preserved ejection fraction: a study of echocardiography versus catheterization. Clin Res Cardiol. 2017 Mar;106(3):192-201. doi: 10.1007/s00392-016-1039-0. Epub 2016 Sep 30. PMID 27695989